CLINICAL TRIAL: NCT01928992
Title: A Multi-reader, Multi-case, Controlled Clinical Trial to Evaluate the Fuji Film 3D Digital Mammography System Used in Conjunction With 2D Digital Mammography in the Detection of Breast Cancer / A Pilot Study
Brief Title: Pilot 3D Mammography Reader Study to Assess Breast Cancer Detection in 3D Versus 2D Digital Mammography
Acronym: 3DM
Status: Completed | Type: Observational
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FMSU2011-003B
Record Dates: First submitted 2013-03-01; First posted 2013-08-27 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
Keywords: Mammography; 3D; Breast Cancer Detection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 3D: Subjects that undergo 3D mammography
  Interventions: Device: 3D
- 2D: Subjects that undergo 2D mammography
  Interventions: Device: 2D

INTERVENTIONS:
Device: 3D — subjects that underwent 3D mammography
  Groups: 3D
Device: 2D — those subjects that underwent 2D mammography
  Groups: 2D

SUMMARY:
The purpose of this pilot study is to provide credible performance estimate information in order to properly plan, design, and power a larger clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects participating in prior FMSU protocol with known clinical status

Exclusion Criteria:

* Subjects with unkown clinical status
* Subjects not truthed in prior FMSU study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with screening and diagnostic 3D or 2D mammography
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Per Breast AUC | 1 Day
  Breast AUC performance metrics to determine if 3D has improved breast cancer detection rate as compared to 2D.

SECONDARY OUTCOMES:
Subject Recall Rate | 1 Day
  For Cancer and Non-Cancer Cases to determine if 3D can reduce the need for follow-up mammography and/or improve time to determination of need for a biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Carl D'Orsi, MD, Principal Investigator — Emory University
Locations (1):
- ACR / Image Metrix, Philadelphia, Pennsylvania, United States